CLINICAL TRIAL: NCT05328505
Title: Molecular Imaging Informed Radiation Dose Escalation to Sites of Recurrent Disease and De-escalation to Uninvolved Areas in Salvage Radiotherapy for Prostate Cancer
Acronym: MIDAS-Prostate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-5147
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; adenocarcinoma; PSMA PET; radical prostatectomy; recurrence
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Recurrence | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Molecular Imaging Informed Radiation Dose Escalation and De-escalation (Experimental): Molecular imaging informed radiation dose escalation to sites of recurrent disease and de-escalation to uninvolved areas.
  Interventions: Radiation: Image-guided Radiotherapy

INTERVENTIONS:
Radiation: Image-guided Radiotherapy — de-escalation radiotherapy to elective volumes + simultaneous integrated boost to PSMA avid lesions delivered in 20 fractions +/- ADT (clinical decision). The elective prostate bed and pelvic lymph node regions will receive 45 Gy. The PSMA-avid lymph node(s) will receive an SIB to 55-60 Gy and/or the PSMA-avid lesion in the prostate bed will receive an SIB to 60 Gy. Pelvic nodal treatment and ADT use will be left to the discretion of the treating physician.

SUMMARY:
This is a Phase II prospective sing-arm trial that is recruiting 60 participants from patients that have biochemical failure after radical prostatectomy with local or regional recurrence proven by PSMA PET. Participants of this study will receive molecular imaging informed radiation dose escalation to site of recurrent disease and de-escalation to uninvolved areas. Participants will be follow-up as per standard of care up to 5 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men older than 18 years old.
* Histologically proven initial diagnosis of adenocarcinoma prostate cancer.
* Previous radical prostatectomy.
* Biochemical relapse with local or regional recurrence proven on PSMA PET.
* Five or less positive nodes on the PSMA PET.
* ECOG 0-1

Exclusion Criteria:

* Presence of para-aortic lymph nodes or distant metastasis.
* Chronic pelvic inflammatory disease.
* Contraindication for radiation treatment.
* Previous radiation treatment within the pelvis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Grade ≥2 Toxicity for GU | Baseline to 5-year follow-up
  Acute (less than or equal to 90 days) toxicity will be evaluated by using prospective follow-up and grading according to the latest version of the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Biochemical Failure Free Survival | Baseline to 5-year follow-up
  Biochemical control rate will be assessed at baseline and at each follow-up visit (1, 3, 6, 12, 18, 24, 36, 48, and 60 months) by the blood level of prostate-specific antigen (PSA) levels
Patient-reported quality-of-life assessed by EPIC-26 | Baseline to 5-year follow-up
  Patient-Reported Quality of Life will be assessed at baseline and at each follow-up visit (3-weeks post intervention then every 6 months until 5 years, or more frequently if clinically necessary) using the following assessment questionnaires: 26-Item Expanded Prostate Cancer Index Composite (EPIC-26)

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No